CLINICAL TRIAL: NCT00240136
Title: Long-term Observation of Patients With Early Rheumatoid Arthritis
Status: Completed | Type: Observational
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Sponsor
Other Study IDs: 91-10-435-32
Record Dates: First submitted 2005-10-13; First posted 2005-10-17 (Estimated); Last update posted 2020-11-17 (Actual); Status verified 2020-11

CONDITIONS: Rheumatoid Arthritis
Keywords: Early, severe
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this research is to observe the effects of RA over a long period in order to learn which of the early characteristics of patients' early RA predict future joint damage and disability. We also investigate whether certain treatments can prevent or slow the development of joint damage and disability. Additionally, the costs and effects of RA on the patient are studied in order to improve the methods used to measure these effects. Clinical, demographic, radiographic, and laboratory measures are taken by the rheumatologist in the office. In addition, patient questionnaires are mailed & completed by the patient and returned to the coordinating center at UCLA. All information obtained by these means will be studied in their effects on early, severe RA.

DETAILED DESCRIPTION:
See Publications

ELIGIBILITY:
Inclusion Criteria:

* >=6 swollen joints & >=9 tender joints
* symmetrical rheumatoid arthritis (RA)
* <= 2 years worth of symptoms
* rheumatoid factor seropositivity

Exclusion Criteria:

* <18 years old
* Inability to see rheumatologist, complete questionnaires (lack of compliance)
* >2 years worth of symptoms

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with rheumatoid arthritis
Sampling Method: Non-Probability Sample
Enrollment: 372 (Actual)
Dates: Start 1993-01; Primary Completion 2020-10-23 (Actual); Study Completion 2020-10-23 (Actual)

PRIMARY OUTCOMES:
Development of joint erosions in the early stages of RA | Baseline, Annual Follow-up
  Measure joint erosions over time

CONTACTS AND LOCATIONS:
Overall Officials: Harold E Paulus, MD, Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA, Los Angeles, California, United States

REFERENCES:
- [Result] Cole JC, Motivala SJ, Khanna D, Lee JY, Paulus HE, Irwin MR. Validation of single-factor structure and scoring protocol for the Health Assessment Questionnaire-Disability Index. Arthritis Rheum. 2005 Aug 15;53(4):536-42. doi: 10.1002/art.21325. PMID 16082630
- [Result] Khanna D, Ranganath VK, Fitzgerald J, Park GS, Altman RD, Elashoff D, Gold RH, Sharp JT, Furst DE, Paulus HE; Western Consortium of Practicing Rheumatologists. Increased radiographic damage scores at the onset of seropositive rheumatoid arthritis in older patients are associated with osteoarthritis of the hands, but not with more rapid progression of damage. Arthritis Rheum. 2005 Aug;52(8):2284-92. doi: 10.1002/art.21221. PMID 16052588
- [Result] Ranganath VK, Elashoff DA, Khanna D, Park G, Peter JB, Paulus HE; Western consortium of practicing rhuemotologists. Age adjustment corrects for apparent differences in erythrocyte sedimentation rate and C-reactive protein values at the onset of seropositive rheumatoid arthritis in younger and older patients. J Rheumatol. 2005 Jun;32(6):1040-2. PMID 15940764
- [Result] Wu H, Khanna D, Park G, Gersuk V, Nepom GT, Wong WK, Paulus HE, Tsao BP. Interaction between RANKL and HLA-DRB1 genotypes may contribute to younger age at onset of seropositive rheumatoid arthritis in an inception cohort. Arthritis Rheum. 2004 Oct;50(10):3093-103. doi: 10.1002/art.20555. PMID 15476205
- [Result] Amjadi S, Khanna D, Park GS, Bulpitt KJ, Wong WK, Paulus HE. Dating the "window of therapeutic opportunity" in early rheumatoid arthritis: accuracy of patient recall of arthritis symptom onset. J Rheumatol. 2004 Sep;31(9):1686-92. PMID 15338485
- [Result] Paulus HE, Oh M, Sharp JT, Gold RH, Wong WK, Park GS, Bulpitt KJ; Western Consortium of Practicing Rheumatologists. Classifying structural joint damage in rheumatoid arthritis as progressive or nonprogressive using a composite definition of joint radiographic change: a preliminary proposal. Arthritis Rheum. 2004 Apr;50(4):1083-96. doi: 10.1002/art.20270. PMID 15077290
- [Result] Paulus HE, Oh M, Sharp JT, Gold RH, Wong WK, Park GS, Bulpitt KJ; Western Consortium of Praticing Rheumatologists. Correlation of single time-point damage scores with observed progression of radiographic damage during the first 6 years of rheumatoid arthritis. J Rheumatol. 2003 Apr;30(4):705-13. PMID 12672187
- [Result] Paulus HE, Wiesner J, Bulpitt KJ, Patnaik M, Law J, Park GS, Wong WK. Autoantibodies in early seropositive rheumatoid arthritis, before and during disease modifying antirheumatic drug treatment. J Rheumatol. 2002 Dec;29(12):2513-20. PMID 12465144
- [Result] Paulus HE, Bulpitt KJ, Ramos B, Park G, Wong WK; Western Consortium of Practicing Rheumatologists. Relative contributions of the components of the American College of Rheumatology 20% criteria for improvement to responder status in patients with early seropositive rheumatoid arthritis. Arthritis Rheum. 2000 Dec;43(12):2743-50. doi: 10.1002/1529-0131(200012)43:123.0.CO;2-A. PMID 11145032
- [Result] Newhall-Perry K, Law NJ, Ramos B, Sterz M, Wong WK, Bulpitt KJ, Park G, Lee M, Clements P, Paulus HE. Direct and indirect costs associated with the onset of seropositive rheumatoid arthritis. Western Consortium of Practicing Rheumatologists. J Rheumatol. 2000 May;27(5):1156-63. PMID 10813281
- [Result] Paulus HE, Ramos B, Wong WK, Ahmed A, Bulpitt K, Park G, Sterz M, Clements P. Equivalence of the acute phase reactants C-reactive protein, plasma viscosity, and Westergren erythrocyte sedimentation rate when used to calculate American College of Rheumatology 20% improvement criteria or the Disease Activity Score in patients with early rheumatoid arthritis. Western Consortium of Practicing Rheumatologists. J Rheumatol. 1999 Nov;26(11):2324-31. PMID 10555885